CLINICAL TRIAL: NCT06133842
Title: CEReBral AutorEgulation in Non-cardiac SuRgery and Relationship to Postoperative DeliriUm State - CERBERUS Trial
Brief Title: CEReBral AutorEgulation in Non-cardiac SuRgery and Relationship to Postoperative DeliriUm State
Acronym: CERBERUS
Status: Recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Samir Kendale, Assistant Professor of Anaesthesia at the Harvard Medical School, Director of Neuroanesthesia at BIDMC, Beth Israel Deaconess Medical Center
Other Study IDs: 2023-P-000843
Record Dates: First submitted 2023-10-17; First posted 2023-11-18 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Perioperative/Postoperative Complications; Postoperative Cognitive Dysfunction; Postoperative Delirium; EEG With Periodic Abnormalities; Intraoperative Hypotension; Cerebral Hypoperfusion
Keywords: EEG; Cerebral Autoregulation; Intraoperative Monitoring
MeSH Terms: conditions — Postoperative Complications; Postoperative Cognitive Complications; Emergence Delirium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Enrolled Participants: Patients above the age of 60 undergoing major non-cardiac surgery requiring invasive MAP monitoring as standard of care. They will be monitored intra-op using non-invasive EEG and CO monitors, which will be correlated with MAP.
  They will also undergo baseline and followup assessment for post-operative delirium using the standardised CAM and MoCA tools administered by study staff.
  Interventions: Diagnostic Test: Intra-op EEG and CO data collection

INTERVENTIONS:
Diagnostic Test: Intra-op EEG and CO data collection — Intra-op EEG and CO data will be collected non-invasively. This will not guide or affect patient care of procedure in any way.
  Other Names: Massimo SEDLINE Root Monitor

SUMMARY:
The goal of this observational study is to learn the how to determine the mean arterial pressure(MAP) or blood pressure level to be maintained during non-cardiac surgery for optimal brain health in patients above the age of 60 undergoing major non-cardiac surgery. The main question[s] it aims to answer are:

* Is there a way to tailor the blood pressure to be maintained in such patients during surgery for optimal brain health using non-invasive monitors that check the brains electrical activity, the electroencephalogram(EEG) monitor, and the brain's blood oxygen levels, the cerebral oximetry(CO) monitor?
* How much does this optimal blood pressure level vary between patients?

Participants will be asked to:

* Complete a questionnaire at the time they enroll into the study, as well as a daily questionnaire to help determine their level of thinking and brain health. This questionnaire will be administered by a member of the study team.
* They will also have an EEG and CO monitoring sticker placed on their foreheads. This will be connected to a monitor that will collect this data just before, during, and after their surgery. The data collected through these monitors will help us with our study goals.

DETAILED DESCRIPTION:
Study Procedures:

Pre-operative:

1. Assessment by an anesthesiologist, and brief patient education about cerebral autoregulation and post-operative delirium.
2. MOCA baseline cognitive assessment by study team member.

Intra-operative:

1. Perioperative EEG Monitoring: EEG stickers will be applied to patient's forehead in pre-op holding area and attached to SedLine Root Monitor (described below in perioperative EEG and Cerebral Oximetry10 (CO) monitoring) at least 5 minutes prior to start of induction.
2. Perioperative CO monitoring: NIRS stickers will be applied to patient's forehead in pre-op holding area and attached to SedLine Root Monitor (described below in perioperative EEG and Cerebral Oximetry (CO) monitoring) at least 5 minutes prior to start of induction.
3. Live collection and processing of data: During surgery, the SedLine Root Monitor (which collects EEG & CO data) and the Operating Room's en-suite Phillips Intellivue monitor (which collects MAP data during surgery) will both be connected to a BIDMC-issued, IS-approved laptop or tablet running the ICM+ software suite. The SedLine Root Monitor and Philips Intellivue Monitor will output their data locally via cables to the system running the ICM+ software suite, which will process and integrate this data in real-time. This processed information will only be collected passively during the surgery, and will not inform or affect clinical care in any way.

   * Perioperative EEG and CO monitoring All patients will undergo EEG and CO monitoring during intraoperative, and possibly the postoperative period (up through 24 hours/until extubation, whichever occurs earlier). The EEG and CO leads will be removed from the patient and monitoring stopped at one of three end-points: a) 24 hours after the end of the surgical procedure b) at time of extubation c) when patient is shifted out of the PACU; whichever comes first. This is to ensure that comprehensive data on cerebral autoregulation during the critical perioperative period is available for any given patient for analysis. Electroencephalograms and CO will be recorded using the SedLine monitor (Masimo Corporation, Irvine California). SedLine is a FDA approved, patient-connected, 4-channel processed electroencephalograph EEG and Cerebral oximetry monitor designed specifically for intraoperative or intensive care use. It displays electrode status, EEG waveforms, Density Spectral Array (DSA) and bilateral regional cerebral oxygen saturation.

The SedLine EEG electrode array records approximately at positions Fp1, Fp2, F7, and F8, with reference approximately 1 cm above Fpz and ground at Fpz. The spectrograms will be computed using the Multitaper method from the unprocessed EEG signals recorded at a sampling frequency of 250 Hz. Individual spectra will be computed in 3-sec windows with 0.5 sec overlap between adjacent windows. Multitaper spectral estimates have near optimal statistical properties that substantially improve the clarity of spectral features.

The CO sensors are applied on the forehead.

* EEG Display The EEG waveforms reflect electrical activity mostly from the front of the brain. The display is configured to contain 4 data input sources, acquired from the 4 sensor electrodes: L1, R1, L2, and R2.

Patient State Index (PSi)31,32 The PSi is a processed EEG parameter that is related to the effect of anesthetic agents, and takes into consideration, among other factors:

1. changes in power in various EEG frequency bands
2. changes in symmetry and synchronization between critical brain regions
3. the inhibition of regions of the frontal cortex.

Density Spectral Array (DSA)31,32 The DSA contains left and right spectrograms representing the power of the EEG on both sides of the brain.

Multitaper DSA32 When using a Multitaper DSA, EEG data are transformed into the frequency domain, which may provide a better display of EEG features.

* Post-operative:

Postoperative pain assessment

Postoperative pain will be assessed with a standard 11-point scale and by pain medication intake. Pain scores will be obtained by asking the subject and also collected from the medical record when documented clinically. Pain medication intake will be extracted from the medical record.

Delirium and cognition assessment Once consent is obtained, a trained research team member will proceed with baseline preoperative and postoperative cognitive, delirium, and depression assessments.

Baseline assessment

This will be conducted by study staff at the time of consent. If the patient cannot complete baseline assessment at time of consent, it may be conducted at a later time before surgery as per the patient's convenience on hospital premises. This will include the assessment of cognitive function using the:

1. Montreal Cognitive Assessment (MoCA)11, supplemented with
2. Days of the week (DOW) & Months of the year (MOY) for additional attention testing
3. Delirium Symptom Interview (DSI) to capture symptoms of delirium
4. Confusion Assessment Method (CAM)12,13: Using data from the cognitive testing and DSI, the researcher will complete the long CAM which includes the diagnosis of delirium using the CAM diagnostic algorithm.

These detailed assessments will take no more than 45 minutes. If this baseline assessment shows a MoCA score <10, the subject will be excluded from the study.

Postoperative assessment On each postoperative day during the hospital stay a research team member will administer a

1. Standard cognitive assessment, including DOW, MOY, CAM, and DSI. These daily assessments will take approximately 10-15 minutes.
2. If a subject is intubated postoperatively, a CAM-ICU will be performed instead of a CAM assessment.
3. If a participant declines to complete a daily standard cognitive assessment, trial staff will offer the 3D-CAM as a shorter alternative. If the participant refuses both the daily standard cognitive assessments and the 3D-CAM, trial staff will use the CAM Only, a conversation-based method to score the CAM.
4. If daily assessments have plateaued for 3 consecutive days (CAM negative each day), they will then only need to be completed every other day, as long as the subject remains CAM negative, until the date of discharge.
5. In addition, medical charts will be reviewed every day until discharge or day 30 (whichever occurs first) to identify delirium. Any events related to delirium during the hospital stay and at the follow-up time points (1 month and 6 months) will be recorded on REDCap eCRF. Events such as trying to get out of bed, verbal abuse, falls, pulling tubes, inappropriate behavior during the hospital stay as noted in the medical charts will be recorded. At phone follow-up: prolonged rehabilitation, cognitive decline will be recorded.

Remote assessments After the patient consents to participate in the study and opts in for phone call assessments, the study team may use the t-MoCA as a substitute to the MoCA for remote assessment of baseline cognition. Additionally, for in-hospital assessments, study investigators may use the a-MoCA as a substitute to the MoCA if an inability for in-person visits arises. Sites may conduct substitution assessments via phone or site-specific HIPAA approved telemedicine video conferencing platform. The a-MoCA and the t-MoCA are identical assessments but differ in naming, where the term "a-MoCA" is used for in-person assessments, and the term "t-MoCA" is used for assessments conducted via phone. Both assessments exclude the visuoconstructional tests of alternating trails, drawing of cube and clock, and animal naming.

Discharge assessment On the day of discharge, the MoCA, with DOW and MOY, the CAM, and the DSI will be completed. (If the discharge assessment was performed in anticipation of discharge on a specific day but the discharge was delayed (i.e., logistical reasons, clinical reasons), this will not be considered a protocol deviation.) If the patient is discharged before a discharge assessment can be done, study staff may contact patient to administer t-MoCA along with DOW and MOY, CAM and DSI.

Follow-up assessment Follow-up assessments will be administered at 1 month (+14 days /- 7 days) and 6 months (+/- 30 days) after the date of surgery. These will be completed by a research team member via telephone and will include a telephone version of the MoCA (t-MoCA), with DOW and MOY, the CAM, SF-12, FRAIL scale, functional activity scale, and long term pain scale and the DSI. These assessments will be done at the patient's convenience and ability to finish the evaluations.

* Delirium treatment The delirium research assessments will not be provided to the treating clinicians. Treating clinicians will assess and treat delirium per the standard of care.
* Data Collection

Patient related information such as baseline characteristics including, comorbid conditions, medications, surgical and anesthetic data will be obtained from Society of Thoracic Surgery database, Anesthesia Information Management Systems and patient's medical record. EEG changes, waveforms and other related data will be recorded from the monitor. Additionally, to track other important factors related to outcome and protocol adherence, study investigators may extract clinical data from the medical record including, but not limited to:

1. Anthropometric data (e.g. age, height, weight, race/ethnicity)
2. Admission type
3. Medications
4. Pain scores
5. Respiratory physiological data
6. Hemodynamic data (e.g. heart rate, blood pressure)
7. Laboratory data
8. Complications data
9. Hospitalization-related time data (e.g. admitting diagnosis, hospital and ICU length of stay)
10. Vital status These data will be merged with subject cognitive assessment data. All data will be stored on password-protected computers, in locked file cabinets and/or offices, or REDCap.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Undergoing any non-cardiac surgeries including but not limited to vascular, hepatobiliary, or complex spine surgeries requiring general anesthesia with arterial catheterization for monitoring

Exclusion Criteria:

1. Non-English speaking (Justification: cognitive assessment instruments are not validated in a sufficient range of languages, and the research team lacks polylingual capabilities or the financial resources to hire interpreters for the duration of all proposed assessments.)
2. Cognitive impairment as defined by total MoCA score < 10 (justification: baseline cognitive dysfunction will confound primary outcome measure)
3. Significant visual impairment (justification: will be difficult for patients to draw individual components in MOCA score)
4. Emergent surgery (justification: insufficient time to initiate intervention)
5. History of stroke within the last 3 months (justification: cognitive dysfunction secondary to stroke can confound outcome measures

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients above the age of 60 scheduled to undergo major non-cardiac surgeries including but not limited to vascular, hepatobiliary, or complex spine surgeries requiring general anesthesia with arterial catheterization for monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
CA state and lower limits of autoregulation (LLA): | 1 week
  The primary outcome will be reliability in the form of an "uptime". This is a calculation of the percentage that each signal provides a feasible measurement, and a percentage that each method of autoregulation calculation produces an output.
  Previous studies have demonstrated a high frequency of uptime, upwards of 90%. CA state and lower limits of autoregulation (LLA) will be calculated using two distinct methods, both previously published and enumerated in the Statistical Consideration section

SECONDARY OUTCOMES:
Duration of burst suppression in EEG | 1 week
  Determine the length of burst suppression on EEG monitoring for each patient. Burst suppression is defined as a period of isoelectric activity in the EEG waveforms.
Incidence of Postoperative Delirium (POD) | Within 1 week
  POD will be diagnosed by our trained research members based on the Confusion Assessment Method (CAM) algorithm postoperatively until discharge.
Cognitive function | 1 month and 6 months
  Postoperative cognitive dysfunction at 1- and 6- months will be assessed with telephone version of the Montreal Cognitive Assessment (t-MoCA) with a maximum positive score of 22. The higher the score, the better the patient's cognitive function.
Hemodynamic stability - Vasopressor Usage | 1 week
  Metrics of total vasopressor dose in norepinephrine equivalents
Hemodynamic stability - Time outside ideal systolic range | 1 week
  Time above/ below 90-130 mmHg systolic blood pressure in minutes
Hemodynamic stability - Area Under Curve | 1 week
  Area under the 65 mmHg mean arterial blood pressure curve in units of mmHg minutes
Hemodynamic stability - Coefficient of Variation recorded as a simple integer | 1 week
  Coefficient of variation of mean arterial blood pressure will be collected from the intraoperative record and medical records to be quantified and compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aries MJ, Czosnyka M, Budohoski KP, Steiner LA, Lavinio A, Kolias AG, Hutchinson PJ, Brady KM, Menon DK, Pickard JD, Smielewski P. Continuous determination of optimal cerebral perfusion pressure in traumatic brain injury. Crit Care Med. 2012 Aug;40(8):2456-63. doi: 10.1097/CCM.0b013e3182514eb6. PMID 22622398
- [Background] Mathieu F, Khellaf A, Ku JC, Donnelly J, Thelin EP, Zeiler FA. Continuous Near-infrared Spectroscopy Monitoring in Adult Traumatic Brain Injury: A Systematic Review. J Neurosurg Anesthesiol. 2020 Oct;32(4):288-299. doi: 10.1097/ANA.0000000000000620. PMID 31306264
- [Background] Hori D, Brown C, Ono M, Rappold T, Sieber F, Gottschalk A, Neufeld KJ, Gottesman R, Adachi H, Hogue CW. Arterial pressure above the upper cerebral autoregulation limit during cardiopulmonary bypass is associated with postoperative delirium. Br J Anaesth. 2014 Dec;113(6):1009-17. doi: 10.1093/bja/aeu319. Epub 2014 Sep 25. PMID 25256545
- [Background] Gaudino M, Rahouma M, Di Mauro M, Yanagawa B, Abouarab A, Demetres M, Di Franco A, Arisha MJ, Ibrahim DA, Baudo M, Girardi LN, Fremes S. Early Versus Delayed Stroke After Cardiac Surgery: A Systematic Review and Meta-Analysis. J Am Heart Assoc. 2019 Jul 2;8(13):e012447. doi: 10.1161/JAHA.119.012447. Epub 2019 Jun 19. PMID 31215306
- [Background] Sun LY, Chung AM, Farkouh ME, van Diepen S, Weinberger J, Bourke M, Ruel M. Defining an Intraoperative Hypotension Threshold in Association with Stroke in Cardiac Surgery. Anesthesiology. 2018 Sep;129(3):440-447. doi: 10.1097/ALN.0000000000002298. PMID 29889106
- [Background] Wachtendorf LJ, Azimaraghi O, Santer P, Linhardt FC, Blank M, Suleiman A, Ahn C, Low YH, Teja B, Kendale SM, Schaefer MS, Houle TT, Pollard RJ, Subramaniam B, Eikermann M, Wongtangman K. Association Between Intraoperative Arterial Hypotension and Postoperative Delirium After Noncardiac Surgery: A Retrospective Multicenter Cohort Study. Anesth Analg. 2022 Apr 1;134(4):822-833. doi: 10.1213/ANE.0000000000005739. PMID 34517389
- [Background] Maheshwari K, Ahuja S, Khanna AK, Mao G, Perez-Protto S, Farag E, Turan A, Kurz A, Sessler DI. Association Between Perioperative Hypotension and Delirium in Postoperative Critically Ill Patients: A Retrospective Cohort Analysis. Anesth Analg. 2020 Mar;130(3):636-643. doi: 10.1213/ANE.0000000000004517. PMID 31725024
- [Background] Whitlock EL, Vannucci A, Avidan MS. Postoperative delirium. Minerva Anestesiol. 2011 Apr;77(4):448-56. PMID 21483389
- [Background] Saczynski JS, Marcantonio ER, Quach L, Fong TG, Gross A, Inouye SK, Jones RN. Cognitive trajectories after postoperative delirium. N Engl J Med. 2012 Jul 5;367(1):30-9. doi: 10.1056/NEJMoa1112923. PMID 22762316
- [Background] Liu X, Akiyoshi K, Nakano M, Brady K, Bush B, Nadkarni R, Venkataraman A, Koehler RC, Lee JK, Hogue CW, Czosnyka M, Smielewski P, Brown CH. Determining Thresholds for Three Indices of Autoregulation to Identify the Lower Limit of Autoregulation During Cardiac Surgery. Crit Care Med. 2021 Apr 1;49(4):650-660. doi: 10.1097/CCM.0000000000004737. PMID 33278074
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Ely EW, Margolin R, Francis J, May L, Truman B, Dittus R, Speroff T, Gautam S, Bernard GR, Inouye SK. Evaluation of delirium in critically ill patients: validation of the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Crit Care Med. 2001 Jul;29(7):1370-9. doi: 10.1097/00003246-200107000-00012. PMID 11445689
- [Background] Montgomery D, Brown C, Hogue CW, Brady K, Nakano M, Nomura Y, Antunes A, Addison PS. Real-Time Intraoperative Determination and Reporting of Cerebral Autoregulation State Using Near-Infrared Spectroscopy. Anesth Analg. 2020 Nov;131(5):1520-1528. doi: 10.1213/ANE.0000000000004614. PMID 33079875
- [Background] Goettel N, Burkhart CS, Rossi A, Cabella BC, Berres M, Monsch AU, Czosnyka M, Steiner LA. Associations Between Impaired Cerebral Blood Flow Autoregulation, Cerebral Oxygenation, and Biomarkers of Brain Injury and Postoperative Cognitive Dysfunction in Elderly Patients After Major Noncardiac Surgery. Anesth Analg. 2017 Mar;124(3):934-942. doi: 10.1213/ANE.0000000000001803. PMID 28151820
- [Background] Chuan A, Short TG, Peng AZY, Wen SYB, Sun AX, Ting TH, Wan AS, Pope L, Jaeger M, Aneman A. Is cerebrovascular autoregulation associated with outcomes after major noncardiac surgery? A prospective observational pilot study. Acta Anaesthesiol Scand. 2019 Jan;63(1):8-17. doi: 10.1111/aas.13223. Epub 2018 Aug 5. PMID 30079514
- [Background] Mol A, Meskers CGM, Sanders ML, Muller M, Maier AB, van Wezel RJA, Claassen JAHR, Elting JWJ. Cerebral autoregulation assessed by near-infrared spectroscopy: validation using transcranial Doppler in patients with controlled hypertension, cognitive impairment and controls. Eur J Appl Physiol. 2021 Aug;121(8):2165-2176. doi: 10.1007/s00421-021-04681-w. Epub 2021 Apr 16. PMID 33860383
- [Background] Manquat E, Ravaux H, Kindermans M, Joachim J, Serrano J, Touchard C, Mateo J, Mebazaa A, Gayat E, Vallee F, Cartailler J. Impact of impaired cerebral blood flow autoregulation on electroencephalogram signals in adults undergoing propofol anaesthesia: a pilot study. BJA Open. 2022 Mar 2;1:100004. doi: 10.1016/j.bjao.2022.100004. eCollection 2022 Mar. PMID 37588691
- [Background] Zhang Y, Tan J, Li P, Zhang X, Yang Y, Liu Y, Fu Q, Cao J, Mi W, Zhang H, Li H. The perioperative application of continuous cerebral autoregulation monitoring for cerebral protection in elderly patients. Ann Palliat Med. 2021 Apr;10(4):4582-4592. doi: 10.21037/apm-21-707. PMID 33966406
- [Background] Burkhart CS, Rossi A, Dell-Kuster S, Gamberini M, Mockli A, Siegemund M, Czosnyka M, Strebel SP, Steiner LA. Effect of age on intraoperative cerebrovascular autoregulation and near-infrared spectroscopy-derived cerebral oxygenation. Br J Anaesth. 2011 Nov;107(5):742-8. doi: 10.1093/bja/aer252. Epub 2011 Aug 10. PMID 21835838
- [Background] Khera T, Mathur PA, Banner-Goodspeed VM, Narayanan S, Mcgourty M, Kelly L, Palihnich K, Novack L, Davis R, Talmor D, Marcantonio ER, Subramaniam B. Scheduled Prophylactic 6-Hourly IV AcetaminopheN to Prevent Postoperative Delirium in Older CaRdiac SurgicAl Patients (PANDORA): protocol for a multicentre randomised controlled trial. BMJ Open. 2021 Mar 10;11(3):e044346. doi: 10.1136/bmjopen-2020-044346. PMID 33692183